CLINICAL TRIAL: NCT07018505
Title: EpCAM-Targeted Surface-Enhanced Raman Spectroscopy Nanotags for Rapid Evaluation of Surgical Margins and Sentinel Lymph Node Metastasis Status in Breast Cancers
Status: Not yet recruiting | Type: Observational
Sponsor: Yunnan Cancer Hospital (Other)
Collaborators: Xiang'an Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Other Study IDs: KYLX2025-149
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Sentinel Lymph Node; Breast Cancers; Metastases; Margin Assessment
Keywords: Sentinel Lymph Node; Surface Enhanced Raman Spectroscopy; EpCAM; Breast cancers; Surgical margin
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Margins of Excision

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surface Enhanced Raman Spectroscopy (SERS) Detection: Intraoperatively, approximately 5 mm samples of tumor and adjacent normal tissues are collected from breast cancer patients after resection. After lymph nodes dissection, the tissues are bisected longitudinally along the maximum cross-section. The collected tissues are then divided into two portions. One portion is weighed, and tissue lysis buffer (RIPA:PIC:PMSF = 100:1:1) is added at a ratio of 5 μL per 1 mg tissue. The tissue is minced into 1 mm fragments on ice, and 3 mm zirconium beads are added for homogenization based on tissue weight. The homogenate is centrifuged at 12,000 g for 2 min at 4°C. The supernatant (50 μL) is collected for detection, and the remaining tissue is reserved for pathological evaluation.
  Interventions: Diagnostic Test: SERS detection

INTERVENTIONS:
Diagnostic Test: SERS detection — Incubation: A mixture of 20 μL (0.5 mg/mL) magnetic beads (MB@RB20115UD), 40 μL SERS nanotags (Au-IR808@RB20115UC), and prepared sample is incubated for 5 min.
  Washing: The supernatant is removed after magnetic separation (30 s), followed by washing with PBST (pH 7.4, 0.05% Tween-20).
  Detection: The separated pellet is resuspended in 10 μL ultrapure water. Then 2 μL solution is spotted onto a 2.5 mm × 2.5 mm gold substrate for air-drying. Raman spectra are acquired using a portable spectrometer (785 nm laser, 500 mW power, 5 s acquisition time, triplicate measurements). Peak areas within 540-570 cm-1 are quantified.

SUMMARY:
For early breast cancer patients, breast-conserving surgery and sentinel lymph node biopsy have emerged as the cornerstone of precision oncology, harmonizing oncologic efficacy with the preservation of breast cosmetics and axillary function. However, conventional margin evaluation relies on subjective experience, leading to positive margin rates of 15%-50% Additionally, sentinel lymph node biopsy faces inherent technical limitations, including prolonged procedural time and significant false-negative rates in detecting micro-metastases. To overcome these challenges, the investigators will introduce a stable "sandwich" EpCAM-targeted surface-enhanced Raman spectroscopy (SERS) detection system to provide rapid evaluation of surgical margins and sentinel lymph node (SLN) metastasis status. In brief, a portion of resected tissue will be immediately homogenized by grinding, and the tissue homogenate will then be analyzed using this detection system to determine its histological characteristics. Pathological confirmation will further validate the method. This approach aims to improve the accuracy and efficiency of intraoperative assessment of breast-conserving surgical margins and SLN status, thereby effectively reducing local recurrence rates and complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between 18-75 years of age
* Female
* Patients presenting with a breast cancer to be resectable on pre-operative assessment
* Good operative candidate
* Subject capable of giving informed consent and participating in the process of consent

Exclusion Criteria:

* Patients unable to participate in the consent process
* Patients had contraindications to surgery, such as serious cardiopulmonary disease, coagulation dysfunction, etc
* Other conditions that the researcher considers inappropriate to participate in the study

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators plan to enroll 40 female patients, aged 18 to 75 years, who have been assessed to have resectable breast cancer and are scheduled to undergo surgery. During the surgery, the resected cancers and lymph nodes will be collected for SERS detection, and Raman signals from the tissues will be collected.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Differentiation of breast cancer and para-cancer tissues as well as metastatic and normal lymph nodes | 1 year
  Raman intensity of breast cancer and para-cancer tissues as well as metastatic and normal lymph nodes after SERS detection.

SECONDARY OUTCOMES:
Expression of EpCAM in the breast cancer and metastatic lymph nodes | 1 year
  Raman intensity of the breast cancer tissues and metastatic lymph nodes with different EpCAM expression level after SERS detection.
The Diagnostic Efficiency of SERS detection | 1 year
  The Area Under the Curve (AUC) of the Receiver Operating Characteristic (ROC), sensitivity and specificity of SERS detection for breast cancers and metastatic lymph nodes.

CONTACTS AND LOCATIONS:
Locations (1):
- Yunnan Cancer Hospital, Kunming, Yunnan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guan PC, Zhang H, Li ZY, Xu SS, Sun M, Tian XM, Ma Z, Lin JS, Gu MM, Wen H, Zhang FL, Zhang YJ, Yu GJ, Yang C, Wang ZX, Song Y, Li JF. Rapid Point-of-Care Assay by SERS Detection of SARS-CoV-2 Virus and Its Variants. Anal Chem. 2022 Dec 27;94(51):17795-17802. doi: 10.1021/acs.analchem.2c03437. Epub 2022 Dec 13. PMID 36511436